CLINICAL TRIAL: NCT02096354
Title: A Phase 2 Randomized, Open-Label Study of RRx-001 vs Regorafenib in Subjects With Metastatic Colorectal Cancer
Acronym: ROCKET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-21-02
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — RRx-001; regorafenib; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RRx-001 followed by irinotecan (Experimental): Once-weekly intravenous RRx-001 at a dose of 4 mg on Days 1, 8, 15, and 22 of a 4-week cycle. On progression and if eligible, patients will receive irinotecan (with or without bevacizumab)
  Interventions: Drug: RRx-001; Drug: Irinotecan
- Regorafenib followed by irinotecan (Active Comparator): Regorafenib daily on Days 1- 21 of a 4-week cycle. On progression and if eligible, patients will receive irinotecan (with or without bevacizumab)
  Interventions: Drug: Regorafenib; Drug: Irinotecan

INTERVENTIONS:
Drug: RRx-001
  Arms: RRx-001 followed by irinotecan
Drug: Regorafenib
  Other Names: Stivarga
  Arms: Regorafenib followed by irinotecan
Drug: Irinotecan — To be dosed after RRx-001 or regorafenib
  Other Names: With or without bevacizumab

SUMMARY:
This two-stage study is designed to compare the safety and activity between RRx-001 against regorafenib followed by irinotecan-based therapies in a parallel comparative study.

Patients who are suffering from advanced or metastatic (meaning the disease has spread) colorectal cancer are invited to participate in this study. There will be two groups of patients (Randomized, open label study), one of these will receive RRx-001 and the other one will receive regorafenib. If patients qualify to participate in this study, they will be randomly assigned to the 'interventional arm' where patients will receive the experimental drug, RRx-001, or the 'control arm' where they will receive the current standard-of-care, Regorafenib. Patients have a 66% chance (2 out of 3) of receiving RRx-001 and a 33 % chance (1 out of 3) of receiving regorafenib.

On progression in the first part of the study, provided ECOG performance status is adequate, and if clinically appropriate i.e. there are no absolute or relative contraindications in the opinion of the Investigator, all subjects will enter the second part of the study and receive irinotecan plus bevacizumab.

Whether patients are given RRx-001 or regorafenib, they will also receive best supportive care, which includes treatments to help manage side effects and symptoms of cancer. This is an open label study, which means patients will know to which of these treatments, RRx-001 or regorafenib, they are assigned.

DETAILED DESCRIPTION:
Purpose This two-stage study is designed to compare the safety and activity between RRx-001 against regorafenib followed by irinotecan-based therapies in a parallel comparative study.

Patients who are suffering from advanced or metastatic (meaning the disease has spread) colorectal cancer are invited to participate in this study. There will be two groups of patients (Randomized, open label study), one of these will receive RRx-001 and the other one will receive regorafenib. Qualifying patients will be randomly assigned (like the flip of a coin) to the 'interventional arm' and receive the experimental drug, RRx-001, or the 'control arm' where they will receive the current standard-of-care, Regorafenib. Patients will have a 66% chance (2 out of 3) of receiving RRx-001 and a 33 % chance (1 out of 3) of receiving regorafenib.

On progression in the first part of the study, provided ECOG performance status is adequate, and if clinically appropriate i.e. there are no absolute or relative contraindications in the opinion of the Investigator, all subjects will enter the second part of the study receive irinotecan plus bevacizumab.

Whether patients are given RRx-001 or regorafenib, they will also receive best supportive care, which includes treatments to help manage side effects and symptoms of cancer. This is an open label study, which means patients will know to which of these treatments, RRx-001 or regorafenib, they are assigned.

Background Oxygen is vital to life, we need it to breathe, for example, but at the same time it gives rise to byproducts that are toxic called free radicals. Free radicals are defined as "oxidants". Similarly, substances that interact with and neutralize free radicals, thus preventing them from causing damage, are called "antioxidants". Examples of recognizable antioxidants are Vitamin E, Vitamin C and beta-carotene. Antioxidants are also known as "free radical scavengers." When free radicals are present in excess of antioxidants damage may occur.

A free radical is an unstable molecule with an unpaired electron, an electrically charged particle, which seeks out another electron to return to a state of balance. An example of a free radical is hydrogen peroxide, recognizable as the household product that "bubbles" when it's poured on wounds. These bubbles come from oxygen free radicals, which are toxic to bacteria and all living cells, including cancer. The fact that these free radicals are toxic has to do with how reactive they are-imagine free radicals as high-speed ball bearings that smash into other molecules in order to "steal" back an electron and end their radical state, which sets off a chain reaction that transforms once stable compounds into a string of reactive radicals.

As new free radicals are created in this chain reaction, they randomly slam into whatever molecules they are closest to and steal their electrons, corroding them, like a biological form of rust. This process is repeated over and over, picking up speed, until an antioxidant can "neutralize" the free radicals and put a stop to the snowball effect. In the same way that this free radical bombardment can damage not only bacteria but also healthy tissues in the body, it is also capable of destroying cancer cells.

The current consensus is that compared to normal tissue tumor cells may accumulate elevated levels of free radicals, which contribute to the development of cancer. This is potentially a fatal weakness, a form of biological "Kryptonite", which can be used to advantage since the addition of even a small amount of free radicals may push the tumor over the edge, past the tipping point, above tolerable thresholds, breaking the camel's back. Similar to the expression "live by the sword, die by the sword", free radicals may lead to the development of cancer but they also are capable of harming it when present in excess.

RRx-001 is a completely new type of drug that comes from the U.S. aerospace or rocket science industry. It is activated to deliver free radicals to tissues that have low levels of oxygen. Compared to normal tissues, which have higher levels of oxygen, most, if not all, tumors exist in a low-oxygen environment, perhaps to prevent oxidation. In this way the free radicals delivered by RRx-001 to cancer cells under low oxygen conditions are able, in theory, to cause their targeted destruction without harming normal cells.

In general, colorectal tumors have low levels of antioxidants and, without this antioxidant protection, these tumors are more likely to be harmed by free radicals, so a treatment like RRx-001, which is able to increase the free radicals in the tumor, may benefit patients with colorectal cancer; this is a reason for studying RRx-001 in colorectal cancer. So far, in a Phase 1 study, 25 men and women with advanced, incurable cancer have received RRx-001 for different lengths of time and at doses that ranged from 10 mg/m2 to 83 mg/m2 once a week.

Regorafenib is a drug approved by the FDA to treat colon cancer after previous chemotherapy is no longer effective. It belongs to a class of targeted drugs known as tyrosine kinase inhibitors. Tyrosine kinases, which play a key role in many cell functions including cell growth and division, are commonly mutated or changed in cancer cells, becoming super-active and producing cells that have uncontrolled growth, and, therefore, blocking them with drugs like regorafenib may keep the cancer cells from growing.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum;
* Subject must have received at least oxaliplatin-, and irinotecan-based regimens with bevacizumab and with, cetuximab or panitumumab if KRAS wildtype and are refractory to irinotecan;
* Subject has measurable disease by radiographic techniques (computerized tomography [CT] or magnetic resonance imaging [MRI]);
* Subjects with a history of brain metastasis are eligible for the study as long as they meet all the following criteria: their brain metastases have been treated, they have no evidence of progression or hemorrhage after treatment, have been off dexamethasone for 4 weeks prior to first study drug administration, and have no ongoing requirement for dexamethasone or anti-epileptic drugs;
* Life expectancy of at least 12 weeks
* Subject's Eastern Cooperative Group (ECOG) performance status is 0 or 1;
* Adequate organ function
* Fertile subjects must use effective contraception during the course of the study and for 30 days following withdrawal from the study;

Exclusion Criteria:

* Clinically significant cardiovascular disease;
* Unresolved toxicity higher attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin- induced neurotoxicity ≤ Grade 2 for at least 14 days;
* Evidence or history of tendency or predisposition to active bleeding. Any hemorrhage or bleeding event of Grade 3 or higher within 4 weeks of start of study medication;
* Symptoms or signs of active brain metastases;
* History of an allergic reaction or intolerance to irinotecan
* Hepatic encephalopathy
* Cholangitis that required treatment or intervention within 4 weeks of study enrollment
* Concurrent anticancer therapy or any cytotoxic therapy within 1 month prior to Day 1. Corticosteroid therapy is not allowed except on dosing days;
* Subject has previously received regorafenib;
* Clear contraindication for systemic corticosteroids (diabetes mellitus is not per se a clear contraindication);
* Severe hypoalbuminemia (albumin < 3.0 g/dL);
* Subjects who are pregnant or lactating or who are planning to become pregnant during the course of the study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-05; Primary Completion 2018-04-13 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, Study Director — EpicentRx, Inc.
Locations (5):
- United States (5):
  - UCSD Moores Cancer Center, La Jolla, California
  - Stanford University, Stanford, California
  - Kaiser Permanete, Honolulu, Hawaii
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Aquilino Cancer Center, Maryland Oncology and Hematology PA, Rockville, Maryland

REFERENCES:
- [Background] Oronsky B, Scribner C, Aggarwal R, Cabrales P. RRx-001 protects normal tissues but not tumors via Nrf2 induction and Bcl-2 inhibition. J Cancer Res Clin Oncol. 2019 Aug;145(8):2045-2050. doi: 10.1007/s00432-019-02958-4. Epub 2019 Jun 27. PMID 31250159
- [Background] Scicinski J, Fisher G, Carter C, Cho-Phan C, Kunz P, Ning S, Knox S, Oronsky B, Caroen S, Parker C, Fanger G, Reid T. The Development Of RRx-001, A Novel Nitric-Oxide-Mediated Epigenetically Active Anticancer Agent. Redox Biol. 2015 Aug;5:422. doi: 10.1016/j.redox.2015.09.035. Epub 2015 Dec 30. PMID 28162292
- [Result] Reid TR, Abrouk N, Caroen S, Oronsky B, Stirn M, Larson C, Beale K, Knox SJ, Fisher G. ROCKET: Phase II Randomized, Active-controlled, Multicenter Trial to Assess the Safety and Efficacy of RRx-001 + Irinotecan vs. Single-agent Regorafenib in Third/Fourth Line Colorectal Cancer. Clin Colorectal Cancer. 2023 Mar;22(1):92-99. doi: 10.1016/j.clcc.2022.11.003. Epub 2022 Dec 2. PMID 36529613
- [Result] Reid T, Dad S, Korn R, Oronsky B, Knox S, Scicinski J. Two Case Reports of Resensitization to Previous Chemotherapy with the Novel Hypoxia-Activated Hypomethylating Anticancer Agent RRx-001 in Metastatic Colorectal Cancer Patients. Case Rep Oncol. 2014 Jan 24;7(1):79-85. doi: 10.1159/000358382. eCollection 2014 Jan. PMID 24575021
- See also: EpicentRx, Inc Home page. — http://www.epicentrx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at four academic medical centers between May 2014 and October 2019. The first participant first visit was May 22, 2014 and the last patient last visit was October 8, 2020.
Pre-assignment Details: 62 participants provided informed consent to participate in the study. Prior to arm assignment, 11 patients dropped out. Thus, 51 participants were eligible to be randomized to a study arm with all 51 receiving treatment on protocol. 34 participants were evaluable and included in the efficacy population within the mITT during the interim analysis. All 51 participants are included in the safety analysis.
Groups:
- Not Randomized: Patients that consented to the study but dropped prior to Randomization.
Period: Overall Study
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan | Not Randomized
Started | 38 | 13 | 11
Completed | 24 | 3 | 0
Not Completed | 14 | 10 | 11
Not completed — Physician Decision | 4 | 5 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Adverse Event | 7 | 4 | 0
Not completed — Ineligible | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Patients consented to the trial but dropped out prior due to ineligibility to proceed to randomization
- Total: Total of all reporting groups
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan | Not Randomized | Total
Number analyzed (Participants) | 38 | 13 | 11 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (10.41) | 61.2 (11.65) | 58.1 (10.25) | 56.4 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 9 | 6 | 36
  Male | 17 | 4 | 5 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 11 | 10 | 42
  Black or African American | 5 | 0 | 0 | 5
  Unknown | 1 | 0 | 1 | 2
  Asian | 11 | 1 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Population: Efficacy Data is analyzed on the 34 patients included in the interim analysis. The team extended the study into a safety extension. All 51 subjects are included in the safety analysis
  participants
    United States: number analyzed (Participants) | 24 | 10 | 11 | 45
    United States | 24 | 10 | 11 | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 47 months
Time Frame: From date of enrollment until death or censorship.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
Number analyzed (Participants) | 24 | 10
months | 8.6 [4.8 to NA] — Based on the Brookmeyer-Crowley CI formula, there is not enough events at the upper limit interval to allow for an estimate, therefore upper limit is NA. | 4.7 [2.2 to NA] — Based on the Brookmeyer-Crowley CI formula, there is not enough events at the upper limit interval to allow for an estimate, therefore upper limit is NA.

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) will be defined as the elapsed time from the from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 77 months
Time Frame: Baseline, every 6-8 weeks while on study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
Number analyzed (Participants) | 24 | 10
months | 6.1 [3.7 to NA] — Based on the Brookmeyer-Crowley CI formula, there is not enough events at the upper limit interval to allow for an estimate, therefore upper limit is NA. | 1.7 [0.7 to NA] — Based on the Brookmeyer-Crowley CI formula, there is not enough events at the upper limit interval to allow for an estimate, therefore upper limit is NA.

3. Secondary Outcome: Number of Adverse Events
Description: Incidence of related Adverse Events (AEs). SAEs and all other non-serious AEs are located in the Reported Adverse Event Module. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 is used to grade adverse events.
Time Frame: Baseline through end of treatment (28 days after last dose of study drug). Approximately 24 weeks.
Measure: Number; unit: Number of total adverse events
Units Other Than Participants: Number of Events
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
Number analyzed (Participants) | 38 | 13
Number analyzed (Number of Events) | 275 | 150
Number of total adverse events
  CTCAE Grade 1 | 184 | 87
  CTCAE Grade 2 | 76 | 48
  CTCAE Grade 3 | 15 | 15
  CTCAE Grade 4 | 0 | 0
  CTCAE Grade 5 | 0 | 0

4. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with ORR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target and non-target disease. PR applied only to participants with at least one measurable lesion. Greater than or equal to 30 % decrease under baseline of the sum of longest diameters of all target measurable lesions.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
Number analyzed (Participants) | 24 | 10
Participants
  Partial Response | 5 | 0
  Stable Disease | 12 | 4
  Progressive Disease | 6 | 6
  Non-Evaluable | 1 | 0

5. Secondary Outcome: Clinical Benefit Rate
Description: The period from study entry through Disease Control. Disease Control Rate (DCR) also correlates to Clinical Benefit Rate (CBR), defined as the percentage of subjects with CR, PR or SD relative to the total number of treated subjects
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
Number analyzed (Participants) | 24 | 10
Participants | 17 | 4

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and **Other (Not Including Serious) Adverse Events** were collected beginning at baseline through end of treatment (28 days after last dose of study drug). All-Cause Mortality was assessed up to 47 months"
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 is used to grade adverse events. Other Adverse Events are reported at 0% or higher for related to study drug RRx-001.
Groups:
- RRx-001 Followed by Irinotecan: Once-weekly intravenous RRx-001 at a dose of 4 mg on Days 1, 8, 15, and 22 of a 4-week cycle. On progression and if eligible, patients will receive irinotecan (with or without bevacizumab)
  RRx-001
  Irinotecan: To be dosed after RRx-001 or regorafenib
- Regorafenib Followed by Irinotecan: Regorafenib daily on Days 1- 21 of a 4-week cycle. On progression and if eligible, patients will receive irinotecan (with or without bevacizumab)
  Regorafenib
  Irinotecan: To be dosed after RRx-001 or regorafenib
Arm/Group | RRx-001 Followed by Irinotecan | Regorafenib Followed by Irinotecan
All-Cause Mortality (participants affected / at risk) | 3/38 | 1/13
Serious Adverse Events (participants affected / at risk) | 14/38 | 7/13
Other Adverse Events (participants affected / at risk) | 19/38 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 Followed by Irinotecan (N=38) | Regorafenib Followed by Irinotecan (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
AV Malformations (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 3 (3) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 Followed by Irinotecan (N=38) | Regorafenib Followed by Irinotecan (N=13)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 6 (7)
Enterovesical fistula (Gastrointestinal disorders) | 2 (8) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (17) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 7 (47) | 2 (2)
Fatigue (General disorders) | 16 (22) | 7 (8)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (11) | 2 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 13 (182) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (7)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (6)
Liver function test abnormal (Investigations) | 2 (8) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (15)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (10) | 0 (0)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (10) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (5) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Palmar-plantar erythrodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Hypertension (Vascular disorders) | 6 (9) | 4 (8)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 2 (2)
Hypercoagulability (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (6) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (16) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (14) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (13) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (14) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (14)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 9 (9)
Headache (Nervous system disorders) | 0 (0) | 6 (7)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02096354/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02096354/ICF_001.pdf